CLINICAL TRIAL: NCT02371486
Title: Does Cesarean Section Scar Defect (Niche) Affect Implantation Rate?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Roy Mashiach, M.D., Vice Chairman Gynecological Department, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-14-1399-RM-CTIL
Record Dates: First submitted 2015-02-10; First posted 2015-02-25 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Infertility; Complications; Cesarean Section
Keywords: cesarean section defect; implantation; ivf
MeSH Terms: conditions — Infertility; Long Qt Syndrome 3 | interventions — Hysteroscopy; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nich Repair (Experimental): Interventions to be administered:
  1. Ultrasound Scan
  2. Diagnostic Hysteroscopy
  3. hysteroscopic repair of cesarean section defect
  4. IVF cycle
  Interventions: Procedure: hysteroscopic repair of cesarean section defect; Procedure: Diagnostic Hysteroscopy; Procedure: Ultrasound Scan; Procedure: IVF Cycle
- No Repair (Sham Comparator): Interventions to be administered:
  1. Ultrasound Scan
  2. Diagnostic Hysteroscopy
  3. IVF cycle Operative hysteroscopy WILL NOT BE PERFORMED
  Interventions: Procedure: Diagnostic Hysteroscopy; Procedure: Ultrasound Scan; Procedure: IVF Cycle

INTERVENTIONS:
Procedure: hysteroscopic repair of cesarean section defect — Operative hysteroscopy for the repair of cesarean section defect is performed under general anesthesia. the cervix is dilated and the cesarean section defect opened. polypoid tissue is ablated
  Other Names: hysteroscopic metroplasty, niche repair
  Arms: Nich Repair
Procedure: Diagnostic Hysteroscopy — Betthochi's method for diagnostic hysteroscopy: No anesthesia will be used. vaginoscopy will be performed, followed by diagnostic hysteroscopy. saline will be used as a distension media. 4.2 mm Storz hysteroscope will be used.
Procedure: Ultrasound Scan — Scanning the uterus with the ultrasound probe . Transvaginal ultrasound usually produces better and clearer images of the female pelvic organs, because the ultrasound probe lies closer to these structures.
  The transvaginal ultrasound probe is thin, about 2cm diameter. The probe is covered with a disposable protective sheath. A small amount of ultrasound gel is placed on the end of this probe. The probe is then gently inserted a short distance into the vagina.
  Other Names: Internal ultrasound
Procedure: IVF Cycle — Controlled ovarian hyperstimulation, followed by Human chorionic Gonadotropin ( hCG) administration, Ovum Pickup and Embryo transfer
  Other Names: IVF Treatment

SUMMARY:
Cesarean scar defects (CSDs), i.e. deficient uterine scars following a cesarean section, involve discontinuity at the site of a previous Cesarean section scar. These anatomical defects have been reported to be associated with postmenstrual spotting, chronic pelvic pain and infertility. Few case series have suggested improved fertility (most probably by improving implantation of embryos) The aim of this study is to prospectively record embryonal implantation rate during IVF in patients with CSDs, and to evaluate the effect of hysteroscopic repair of CSDs on fetal implantation during IVF.

DETAILED DESCRIPTION:
150 patients undergoing IVF after cesarean section will be recruited. demographic, clinical and treatment data will be collected. ultrasound and hysteroscopic evaluation of the CSD will be performed. IVF treatment will be provided. In case of failure of IVF treatment, patients will be randomized to hysteroscopic repair of CSD versus second IVF treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing IVF after cesarean section

Exclusion Criteria:

* Patients who underwent CSD repair
* Patients with low ovarian reserve
* Patients with hydrosalpinges, endometriosis, adenomyosis, submucous fibroids or polyps

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Embryo implantation rate | completion of two IVF cycles after randomization - approx. 2 months
  Embryo implantation rate during IVF

SECONDARY OUTCOMES:
Fluid in Uterus | completion of two IVF cycles after randomization - approx. 2 months
  Detection of fluid in the uterine cavity during menotropin stimulation in IVF treatment
Correlation between size and type of the defect fluid accumulation | completion of two IVF cycles after randomization - approx. 2 months
  Correlation between the size and type of the defect and the detection of fluid in the uterine cavity during menotropin stimulation in IVF treatment
Correlation between the size and type of the defect and implantation rate during IVF treatment | completion of two IVF cycles after randomization - approx. 2 months
  Correlation between the size and type of the defect and implantation rate during IVF treatment

CONTACTS AND LOCATIONS:
Locations (1):
- The chaim sheba medical center,Tel Hashomer, Ramat Gan, Israel